### Statistical Analysis Plan

A double-blinded, randomized, placebo-controlled, parallel-group study evaluating the effect of the probiotic *Lactobacillus reuteri* on recurrent urinary tract infection (UTI) in adult women recently treated for UTI.

Sponsors study code: CSUB0144

NCT 03366077

Document Date: 3 sept 2019



CTC Project Code: 2017-149

### CONFIDENTIAL

### Statistical Analysis Plan (SAP)

| Sponsor: | BioGaia AB |
|---|---|
| Study code: | BioGaia CSUB 0144 |
| Study title: | A double-blinded, randomized, placebo-<br>controlled, parallel-group study evaluating<br>the effect of the<br>probiotic <i>Lactobacillus reuteri</i> on recurrent<br>urinary tract infection (UTI) in adult<br>women recently<br>treated for UTI. |
| Date: | 27MAR2019 - Draft 1<br>08AUG2019 - Final 1.0<br>03SEP2019 - Final 2.0 |

CTC Project Code: 2017-149

| 1 | VER | RSION HISTORY | 4 |
|---|----------------|--------------------------------------------------|------|
| 2 | INT | RODUCTION | 4 |
| 3 | | NICAL STUDY DETAILS | |
| | 3.1 | Clinical Study Objectives and Endpoints | |
| | 3.2 | Clinical Study Design | |
| | 3.3 | Statistical Hypotheses | |
| | 3.4 | Number of Subjects | |
| | 3.5 | Methods of Assigning Subject to IMP | |
| | 3.6 | Blinding | |
| 4 | | TISTICAL AND ANALYTICAL PLANS | |
| | 4.1 | Sample Size Determination | |
| | 4.2 | Definition of Analysis Sets | |
| | 4.2.1 | | |
| | 4.2.2 | | |
| | 4.2.3 | | |
| | 4.3 | Definition of Baseline | |
| | 4.4 | Summary Statistics | |
| | 4.5 | Significance Level | |
| | 4.6 | Multiple Comparisons/Multiplicity | |
| | 4.7 | Handling of Drop-outs, Missing Data and Outliers | |
| | 4.8 | Adjustment for Covariates | |
| | 4.9 | Multicentre Studies | |
| | 4.10 | Examination of Subgroups | |
| | 4.11 | Blind Review | |
| | 4.12 | Deriving of confirmed and unique UTI | |
| 5 | <b>SUB</b> 5.1 | Subject Disposition | |
| | 5.2 | Baseline Characteristics and Demographics | |
| 6 | | ATMENT INFORMATION AND EXTENT OF EXPOSURE | |
| U | 6.1 | Active Treatment | |
| | 6.2 | Prior and Concomitant Medications | .13 |
| 7 | STA | TISTICAL METHODOLOGY | 14 |
| | 7.1 | Primary endpoint(s) Analysis | |
| | 7.1.1 | Main analytical approach | . 14 |
| | 7.1.2 | Sensitivity analysis | . 14 |
| | 7.1.3 | Supplementary analyses | . 14 |
| | 7.1.4 | Presentation | . 14 |
| | 7.2 | Secondary Endpoint(s) Analysis | .14 |



CTC Project Code: 2017-149

| | 7. | .2.1 | Definition of endpoint(s) | 14 |
|---|---|---|---|---|
| | 7. | .2.2 | Analysis safety endpoint(s) | 15 |
| | 7. | .2.3 | Main analytical approach | 15 |
| | 7. | 2.4 | Sensitivity analysis | 15 |
| | 7. | 2.5 | Supplementary analyses | 15 |
| | 7. | 2.6 | Presentation | 15 |
| | 7.3 | Tert | iary/Exploratory Endpoint(s) Analysis | 15 |
| | 7.4 | Disc | ontinuation | 15 |
| | 7.5 | Othe | er Analyses | 15 |
| | 7.6 | Inte | rim Analysis | 15 |
| 8 | CI | HANGE | S FROM THE CSP | 16 |
| 9 | ST | <b>TATIS</b> 1 | TICAL DELIVERABLES | 17 |
| 10 | ) | SOFT | VARE | 18 |
| 11 | - | APPR | OVAL | 19 |
| 11<br>12 | | | DRTIVE DOCUMENTATION | |
| 12 | | SUPPO | | 20 |
| 12 | , | SUPP( | DRTIVE DOCUMENTATION | <b>20</b><br>20 |
| 12<br>13 | 12.1<br>12.2 | SUPPO<br>Appo<br>Appo<br>DEMO | PRTIVE DOCUMENTATIONendix 1. – List of Abbreviationsendix 2. – Changes to Protocol-Planned Analyses | 20<br>20<br>20<br>21 |
| 12<br>13 | 12.1<br>12.2 | Appe<br>Appe<br>DEMO<br>Dem | ORTIVE DOCUMENTATION endix 1. – List of Abbreviations endix 2. – Changes to Protocol-Planned Analyses GRAPHIC DATA lographic information | 20<br>20<br>20<br>21<br>21 |
| 12<br>13 | 12.1<br>12.2 | Appe<br>Appe<br>DEMO<br>Dem | PRTIVE DOCUMENTATIONendix 1. – List of Abbreviationsendix 2. – Changes to Protocol-Planned Analyses | 20<br>20<br>20<br>21<br>21 |
| 12<br>13 | 12.1<br>12.2<br>13.1 | Appo<br>Appo<br>Appo<br>DEMO<br>Dem<br>Med | ORTIVE DOCUMENTATION endix 1. – List of Abbreviations endix 2. – Changes to Protocol-Planned Analyses GRAPHIC DATA lographic information | 20<br>20<br>20<br>21<br>21<br>22 |
| 12<br>13 | 12.1<br>12.2<br>13.1<br>13.2 | Appo<br>Appo<br>Appo<br>DEMO<br>Dem<br>Med<br>Subj | ORTIVE DOCUMENTATION endix 1. – List of Abbreviations endix 2. – Changes to Protocol-Planned Analyses GRAPHIC DATA lographic information ical/Surgical history | 20<br>20<br>20<br>21<br>21<br>22<br>23 |
| 12<br>13 | 12.1<br>12.2<br>13.1<br>13.2<br>13.3 | Appo<br>Appo<br>DEMO<br>Dem<br>Med<br>Subj | PRTIVE DOCUMENTATION endix 1. – List of Abbreviations endix 2. – Changes to Protocol-Planned Analyses GRAPHIC DATA lographic information ical/Surgical history ect disposition and exposure | 20<br>20<br>20<br>21<br>21<br>22<br>23<br>24 |
| 13 | 12.1<br>12.2<br>13.1<br>13.2<br>13.3 | SUPPO<br>Appo<br>Appo<br>DEMO<br>Dem<br>Med<br>Subj<br>CON<br>Prim | ORTIVE DOCUMENTATION endix 1. – List of Abbreviations endix 2. – Changes to Protocol-Planned Analyses GRAPHIC DATA ographic information ical/Surgical history ect disposition and exposure COMITANT MEDICATIONS | 20<br>20<br>20<br>21<br>21<br>22<br>23<br>24<br>25 |
| 13 | 12.1<br>12.2<br>13.1<br>13.2<br>13.3<br>13.4 | SUPPO<br>Appo<br>Appo<br>DEMO<br>Dem<br>Med<br>Subj<br>CON<br>Prim | PRTIVE DOCUMENTATION endix 1. – List of Abbreviations endix 2. – Changes to Protocol-Planned Analyses GRAPHIC DATA ographic information ical/Surgical history ect disposition and exposure COMITANT MEDICATIONS ary Endpoint: XXXX | 20<br>20<br>20<br>21<br>21<br>22<br>23<br>24<br>25<br>26 |
| 13 | 12.1<br>12.2<br>13.1<br>13.2<br>13.3<br>13.4<br>13.5 | SUPPO<br>Appo<br>Appo<br>Dem<br>Dem<br>Med<br>Subj<br>CON<br>Prim<br>Cont | PRTIVE DOCUMENTATION endix 1. – List of Abbreviations endix 2. – Changes to Protocol-Planned Analyses GRAPHIC DATA ographic information ical/Surgical history ect disposition and exposure COMITANT MEDICATIONS ary Endpoint: XXXX inuous variables measured over time | 20<br>20<br>20<br>21<br>21<br>22<br>23<br>24<br>25<br>26<br>27 |



CTC Project Code: 2017-149

### 1 VERSION HISTORY

This Statistical Analysis Plan (SAP) for study BioGaia CSUB 0144 is based on the protocol dated 24OCT2017.

**Table 1 SAP Version History Summary** 

| SAP<br>version | Approval<br>Date | Changes | Rationale |
|----------------|------------------|---------|------------------|
| 1 | 08AUG2019 | NA | Original version |
| 2 | xxAUG2019 | | |

### 2 INTRODUCTION

This Statistical Analysis Plan (SAP) gives details regarding the statistical analyses and data presentation outlined in the final Clinical study protocol (CSP) for the study BioGaia CSUB 0144. Any changes from the final CSP are given in Section 0.



CTC Project Code: 2017-149

### **3 CLINICAL STUDY DETAILS**

### 3.1 Clinical Study Objectives and Endpoints

| Objects | Estimands/Endpoints |
|---|---|
| Primary | |
| The primary objective is to evaluate the effect of oral supplementation with Lactobacillus reuteri on the frequency of confirmed UTI during six months from start of intervention in adult women with recurrent UTI. | <ul> <li>Mean number of confirmed UTIs<br/>during six months from start to<br/>intervention, as compared to placebo.</li> </ul> |
| Secondary | |
| <ul> <li>To evaluate the effect of oral supplementation with Lactobacillus reuteri on the frequency of confirmed UTI during the three months' intervention period and during the three months' follow-up period, respectively.</li> <li>To evaluate the effect of oral supplementation with Lactobacillus reuteri on time to first relapse of UTI.</li> <li>To evaluate the effect of oral supplementation with Lactobacillus reuteri on relapse rate at three and six months after start of intervention.</li> <li>To assess the tolerability of oral supplementation with Lactobacillus reuteri in adult women with recurrent UTI.</li> </ul> | <ul> <li>Mean number of confirmed UTIs during the three months' intervention period, as compared to placebo.</li> <li>Mean number of confirmed UTIs during the three months' follow-up period, as compared to placebo.</li> <li>Mean time from start of intervention to first relapse of UTI, as compared to placebo.</li> <li>Proportion of subjects (%) who experienced at least one confirmed UTI during three months from start of interventions, as compared to placebo.</li> <li>Proportion of subjects (%) who experience at least one confirmed UTI during six months from start of intervention, as compared to placebo.</li> <li>Occurrence and frequency of Adverse Events (AEs)</li> </ul> |
| Tertiary/Exploratory | |
| Not applicable | Not applicable |

| Objective (Initial Grategory) Statistical Endocation (Initial Grategory) Statistical Endocation (Initial Grategory) Population (Initial Grategory) Profit (Initial Grategory) Pro | | | Estimand <sup>1</sup> | 3 | | |
|---|---|---|---|---|---|---|
| Chinds Category Category Endpoint Population IES¹ Introduction Ites¹ Primary Objective: To compare the efficacy superiority of the probiotic Lactobacillus reuter it to placebo/active control in participants of adult women with the frequency of performance of UTI Change from baseline in FAS Initiation of rescue Mean difference between initiation of rescue New episode of UTI Primary/MACP Change from baseline in Introduction of the end six months. Initiation of rescue Initiation of rescue Initiation of rescue New episode of UTI Primary/MACP Change from baseline in Introduction of three and six months. Initiation of rescue Initiation of rescue Initiation of rescue Sensitivity Sensitivity Introduction of tree and six months. Internet to six months. Internet to six months. Supplementary Number of confirmed UTI FAS Captured in variable of three to six months. Internet to six months. Number of confirmed Secondary/MCP Accondary/MCP | Objective | Statistical | Variable/ | | | PLS1 |
| Primary Objective: To compare the efficacy superiority of the probiotic Lactobacillus reuter to placebo/active control in participants of adult women with the frequency of confirmed UTI. New episode of UTI. New episode of UTI. Primary/MCP Sensitivity Sensitivity Supplementary Number of confirmed UTI. Supplementary Number of confirmed UTI. Secondary/MCP Number of confirmed UTI. Secondary/MCP Number of confirmed UTI. Secondary/MCP Number of confirmed UTI. Secondary/MCP Number of confirmed UTI. Time from stat of legistic regression) Time from stat of legistic regression Time from telapse Exploratory Time from to relapse Exploratory Time from stat of legistic regression Time from time from stat of legistic regression Time from time from stat of legistic regression Time from time f | Clinical Category | Category | Endpoint | Population | IES¹ | (Analysis) |
| pisode of UTI Primary/MCP Change from baseline in at three and six months. Sensitivity Supplementary Supplementary Secondary/MCP Secondary Sec | Primary Objective: To co confirmed UTI. | mpare the efficacy su | periority of the probiotic Lact | obacillus reuteri to placeb | o/active control in participants | of adult women with the frequency of |
| sensitivity Supplementary Supplementary For scondary/MCP Secondary For striany In unamber of confirmed UTI Secondary To mumber of confirmed UTI FAS Testument to intervention Gatherent to intervention FAS Medication: "had rescue medication not been initiated" (hypothetical). Discontinuation of treatment due to adverse event (AE): "regardless of treatment due to adverse event (AE): "regardless of treatment due to deferse policy) Testument adverse adherent to intervention FAS Testinary Testument intervention FAS Tertiary Tertiary Testument to intervention FAS Tertiary Tertiary Testument of intervention FAS Tertiary Testument of intervention FAS Tertiary Testument of intervention Testument to intervention FAS Tertiary Testument of intervention Testument to relapse Testument and testument to intervention Testument and testument to intervention Testument and testument and testument to intervention Testument and testument and tes | New episode of UTI | Primary/MCP | Change from baseline in | FAS | Initiation of rescue | Mean difference between |
| sensitivity Sensitivity Supplementary Number of confirmed UTI Secondary/MCP Secondary Tom start of Tertinary Tom start of Tertinary T | | | number of confirmed UTI | | medication: "had rescue | interventions |
| Sensitivity Sensitivity Supplementary Supple | | | at three and six months. | | medication not been | (LSMD from CFB ANCOVA with MI |
| Sensitivity Sensitivity Supplementary Supplementary Number of confirmed UTI FAS Execondary/MCP Secondary/MCP Secondary Tom start of Tertiary Tom start of Tertiary Transport (Composite) Tertiary Tertiar | | | | | initiated" (hypothetical). | from participants from same |
| Sensitivity Supplementary Supplementary Number of confirmed UTI FAS rescondary/MCP Secondary/MCP Secondary Teertiary Supplement to intervention of adherent to intervent to in | | | | | | randomized arm off-treatment at |
| Sensitivity Sensitivity Supplementary Initiated at three and six months and remained adherent to intervention Secondary/MCP Secondary/MCP Secondary Textiary Secondary Sec | | | | | Discontinuation of | three to six months) |
| Sensitivity Supplementary Supp | | | | | treatment due to adverse | |
| Supplementary Number of confirmed UTI responder (criterion) and rescue medication not initiated at three and six months and remained adherent to intervention FAS Captured in variable definition (composite) er of confirmed Secondary/MCP Adherent to intervention FAS Association (composite) from start of Tertiary FAS Association rendion to relapse Exploratory Exploratory Association | | Sensitivity | | | event (AE): "regardless of | (LSMD from CFB ANCOVA with |
| Supplementary Number of confirmed UTI FAS Captured in variable responder (criterion) and resound responder (criterion) and rescue medication not initiated at three and six months and remained adherent to intervention adherent to intervention for Secondary Secondary Secondary Tertiary FAS Captured in variable adjinition (composite) FAS AS BEAS Condary Tertiary FAS Cond | | | | | treatment discontinuation | reference-based MI) |
| Supplementary Number of confirmed UTI FAS Captured in variable responder (criterion) and rescue medication not initiated at three and six months and remained adherent to intervention Secondary/MCP FAS adherent to intervention FAS condary Secondary Secondar | | | | | due to AE" (treatment | |
| Supplementary Number of confirmed UTI FAS Captured in variable responder (criterion) and responder (criterion) and rescue medication not initiated at three and six months and remained adherent to intervention ser of confirmed Secondary/MCP FAS Exploratory Tom start of Tertiary FAS Tertiary FAS Tertiary Fastors FAS Tertiary FAS TERTIAL TERTI | | | | | policy) | |
| er of confirmed Secondary/MCP Secondary Second | | Supplementary | Number of confirmed UTI | FAS | Captured in variable | Odds ratio between interventions |
| rescue medication not initiated at three and six months and remained adherent to intervention Secondary/MCP adherent to intervention Secondary rom start of Tertiary rom start of Exp.'oratory ention to relapse Exp.'oratory | | | responder (criterion) and | | definition (composite) | (Logistic regression) |
| er of confirmed Secondary/MCP adherent to intervention secondary rom start of Tertiary Exp.'oratory initiated at three and six months and remained adherent to intervention adherent to intervention Secondary Tertiary Tertiary Exp.'oratory | | | rescue medication not | | | |
| er of confirmed Secondary/MCP adherent to intervention adherent to intervention secondary From start of Tertiary Exp.loratory Tertiary Exp.loratory | | | initiated at three and six | | | |
| er of confirmed Secondary/MCP adherent to intervention Secondary rom start of Tertiary ention to relapse Exp.oratory | | | months and remained | | | |
| er of confirmed Secondary rom start of Tertiary ention to relapse Exploratory | | | adherent to intervention | | | |
| er of confirmed rom start of ention to relapse | | Secondary/MCP | | FAS | | |
| rom start of<br>ention to relapse | Number of confirmed | Secondary | | | | |
| rom start of<br>ention to relapse | UTI | | | | | |
| ention to relapse | Time from start of | Tertiary | | | | |
| of UT! | intervention to relapse | Exp!oratory | | | | |
| | of UTI | | | | | |
| | period and during the three months' follow-up period, respectively. | ree months' follow-up | period, respectively. | | | |

Protocol Number: BioGaia CSUB 0144 CTC Project Code: 2017-149

| | | Estimand <sup>1</sup> | | | |
|---|---|---|---|---|---|
| Objective | Statistical | Variable/ | | | PLS <sup>1</sup> |
| Clinical Category | Category | Endpoint | Population | IES1 | (Analysis) |
| 2. To evaluate the effect α | of oral supplementat | 2. To evaluate the effect of oral supplementation with Lactobacillus reuteri on time to first relapse of UTI. | on time to first relapse of l | JTI. | |
| 3. To evaluate the effect α | of oral supplementat | ion with Lactobacillus reuteri | on relapse rate at three an | 3. To evaluate the effect of oral supplementation with Lactobacillus reuteri on relapse rate at three and six months after start of intervention. | rvention. |
| 4. To assess the tolerabili | ty of oral supplemen. | 4. To assess the tolerability of oral supplementation with Lactobacillus reuteri in adult women with recurrent UTI. | eri in adult women with rec | current UTI. | |
| AEs | | Presence of TEAEs | Safety | | Record from start of IP intervention. |
| | | | Safety | | Medical events occurring between |
| | | | | | screening and start of IP |
| | | | | | intervention. |
| SAEs | | | Safety | | Record from start of IP intervention. |
| | | | Safety | | Medical events occurring between |
| | | | | | screening and start of IP |
| | | | | | intervention. |

IES = Intercurrent event(s) strategy; PLS = Population-level summary.

CFB = Change From Baseline

LSMD = Least Squares Mean Difference

FAS = Full Analysis Set

TEAE = Treatment Emergent Adverse Event

MCP = Multiple comparisons procedure: FWER controlled for hypothesis testing of selected endpoints as specified in Section <cross-reference>.

<sup>1</sup> All estimand attributes explicitly identified for primary/secondary and selected key estimands only.



CTC Project Code: 2017-149

### 3.2 Clinical Study Design

A double-blinded, randomized, placebo-controlled, parallel-group study.

The study will be performed in female subjects aged 18-50 since this is the population expected to benefit from the intervention studied.

The study structure based on assessments using video -and phone-calls to ensure access to a broad population in a wide area although only one study site will be involved.

No clinical safety assessments are considered necessary considering the general good safety profile of probiotics.

### 3.3 Statistical Hypotheses

Hypothesis:

 $H_0$ : Mean number of UTIs in Probiotic group = Mean number of UTIs in the placebo group.

H₁: Mean number of UTIs in Probiotic group ≠ Mean number of UTIs in the placebo group.

### 3.4 Number of Subjects

The number of subjects needed to verity that the mean number of UTIs during six months for the probiotic will be 0.75 and for placebo 1.35 with a common standard deviation of 1.15, will be 118 (1:1 randomization) using a significance level of 5% and a power of 80%.

Assuming a drop-out rate of 15% a total of 140 subjects will be included, 70 in each intervention arm

### 3.5 Methods of Assigning Subject to IMP

The study will consist of a combined screening and randomization assessment, an IP first dose confirmation call and monthly follow up assessments for six months. The screening and randomization assessment will be performed as a phone call or a video-call using an e-health digital platform. Informed consent will be signed via Bank ID. The monthly follow-up assessments will be performed either as a video-call or by phone. However, physical visits to the clinic at CTC AB might be performed for subjects in Uppsala.

Subjects will be recruited from advertising (e.g in social media, at pharmacies etc.). The subjects will contact the study site by phone or e-mail. Brief oral information about the study will be given and pre-defined pre-screening questions will be asked. Written information will be sent to the subjects qualified for screening together with instructions regarding the e-health platform and Bank ID signing procedures.

During the screening and randomization assessment, full information about the study will be given and informed consent. Information regarding demographics, weight, height, medical history, UTI history, medication history, use of restricted products, and pregnancy will be collected and diet restrictions. Subjects will be screened for eligibility as per the pre-defined eligibility criteria.

Eligible and consenting subjects will be randomized to intervention with either *Lactobacillus reuteri* or placebo. The subject will be provided with Investigational Product (IP) for three months (90 days) and niture/Leu urine test kits. Instructions to start intake of IP as soon as the IP has been picked-up will be given. The subject will be contacted by study staff 1-3 days after randomization to confirm that first IP dose has been taken.

At the monthly assessments (video-call/phone-call or visit), the subject will be asked to answer predefined questions regarding symptoms (frequency, urgency and dysuria). If two out of three symptoms are present a UTI is confirmed. If only one symptom is present the subject will perform a niture/Leu urine test at home, preferably on urine retained in the bladder for approximately 3 hrs. If the test is positive (one of two analyses), a UTI is confirmed and the subject is recommended to contact the health care system for consultation regarding antibiotic treatment. Information on AEs, concomitant medications, use of restricted products, pregnancy, and compliance with instructions for IP intake will be collected.



CTC Project Code: 2017-149

An electronic diary will be used by the subject during the study period for recording of occurrence of UTI symptoms and sexual activity (frequency of intercourse, new partner, use of condom with spermicide).

The monthly follow-up assessment after six months will be the final study assessment. Number of empty sachets and any unused IP will be reported to CTC AB by the subject and documented by site staff on the IP accountability list.

### 3.6 Blinding

This is a double-blinded study. All study staff, including the Principal Investigator and the persons performing the subject assessments using the video link or phone calls, will be blinded during the study. Sealed individual treatment code envelopes will be kept at the clinic to be able to break the code if any emergency occurs, as judged by the Investigator.



CTC Project Code: 2017-149

### 4 STATISTICAL AND ANALYTICAL PLANS

### 4.1 Sample Size Determination

A total of 140 subjects completed will be required, 70 in each intervention arm.

### 4.2 Definition of Analysis Sets

### 4.2.1 Full Analysis Set

The Full Analysis Set (FAS) will consist of all subjects who have been randomized and received at least one dose of Intervention.

### 4.2.2 Per Protocol Analysis Set

The Per Protocol Set (PPS) will consist of all subjects who have been randomized, completed the three months of intervention period and without any major protocol deviations. All deviations will be presented and discussed at the clean file meeting. If the compliance with the IP regimen should be below 80% the subject will not be included in the PPS population. The definition of compliance by calculating the number of days in the study (90 days) in relation to number of unused IP as reported by the subject.

$$\frac{90 \ days - number \ of \ doses \ unused}{study \ length \ with \ a \ maximum \ of \ 90 \ days} \geq 0.80$$

Calculations for compliance will be used on visit 4 (3 month).

Subjects who have been used prohibited medications, long term antibiotics or Hipex during the study will be excluded from PPS.

Subjects not participated at visit 4 and 7 (3 month and 6 month) will not be included in the PPS population.

### 4.2.3 Use of analysis set

The FAS population will be used for both of efficacy (primary objectives and secondary objectives) and safety evaluation and the PPS will only be used for the efficacy (i.e. secondary objectives) evaluations.

### 4.3 Definition of Baseline

Baseline measurement is defined as the latest measurement prior to first dose of IMP.

### 4.4 Summary Statistics

In general, all data collected will be presented with summary statistics and given in patient data listings. Summary statistics will include at least number of patients, mean, standard deviation, median, minimum and maximum for continuous data and frequency and percentage for categorical data. Table with summary statistics will be divided by treatment group and dose group, and visit where applicable. Patient data listings will be sorted by treatment, subject and timing of assessments.

### 4.5 Significance Level

The estimated intervention difference will be presented by LSMeans and a 95% confidence interval.

### 4.6 Multiple Comparisons/Multiplicity

All statistical significant findings need to be interpreted from a medical perspective and judged as clinical relevant or not and therefore no adjustment for multiplicity will be performed.



CTC Project Code: 2017-149

### 4.7 Handling of Drop-outs, Missing Data and Outliers

Outliers will be included in summary tables and listings, and will not be handled separately in any analyses. No imputation of data will be performed.

### 4.8 Adjustment for Covariates

History of UTIs and age will be used as covariates in the analysis of mean number of UTIs. Sexual activity will only be used as a covariate in the analysis if it is possible.

### 4.9 Multicentre Studies

No adjustment for centre will be applied, since this will not be considered as a multi-centre study.

### 4.10 Examination of Subgroups

Will be discussed with the client.

### 4.11 Blind Review

Not applicable.

### 4.12 Deriving of confirmed and unique UTI

Definitions of confirmed UTI – If a subject have at least one of three statements:

- A total number of symptoms ≥ 2
- A positive urine test registered at site
- A positive test, self-reported

Definitions of unique UTI – If a subject have no confirmed UTIs within 14 days prior to the current confirmed UTI and have at least one of two statements:

- Confirmed UTI registered at site
- Confirmed UTI, self-reported and no confirmed self-reported UTIs within 14 days prior to the UTI (only applied to self-reported UTIs, since UTIs registered at site are assigned the date of telephone contact and not the date of the actual UTI)

Assigning dates to confirmed UTIs reported by site personnel: Date of previous telephone contact used if date is  $\leq$  14 days prior to registering in the UTI log. In case of later reporting of UTIs, the closest unmatched event date with indication of UTI prior to registration is used as date.



CTC Project Code: 2017-149

### **5 SUBJECTS**

### 5.1 Subject Disposition

The number of subjects that entered the study, withdrawn subjects, completed subjects and the number of subjects at each visit will be summarized by treatment.

### **5.2 Baseline Characteristics and Demographics**

The following baseline characteristics will be given by treatment:

- Age
- Ethnicity
- Weight, height and BMI
- Medical/Surgical history
- UTI history



CTC Project Code: 2017-149

### 6 TREATMENT INFORMATION AND EXTENT OF EXPOSURE

### **6.1 Active Treatment**

The number of subjects on each IP will be tabulated with start time, stop time and duration of application will be tabulated using listings and summary statistics.

### **6.2 Prior and Concomitant Medications**

Prior and concomitant medication data will be listed and tabulated by ATC code. Prior and concomitant medications will be coded according to the World Health Organization (WHO) Anatomic Therapeutic Chemical (ATC) classification system.



CTC Project Code: 2017-149

### 7 STATISTICAL METHODOLOGY

All parameters will be presented by treatment and visit using summary statistics. Additional statistical analyses are specified below.

### 7.1 Primary endpoint(s) Analysis

The primary endpoint will be the mean number of confirmed UTIs during six months from start of intervention, as compared to placebo.

The mean number of UTIs per intervention group will be estimated based on the total number of UTIs by subject.

An additional analysis will be made to include the subjects who have been used prohibited medications, long term antibiotics and Hiprex during the study.

### 7.1.1 Main analytical approach

The mean number of UTIs will be analysed using analysis of covariance with intervention, UTI history and age as independent variables. Sexual activity will only be used in the analysis if it is possible.

### 7.1.2 Sensitivity analysis

No sensitivity analysis for primary endpoint(s) will be performed.

### 7.1.3 Supplementary analyses

No supplementary analysis for primary endpoint(s) will be performed.

### 7.1.4 Presentation

All graphs and tables will be presented in demographic data, section 13.

### 7.2 Secondary Endpoint(s) Analysis

### 7.2.1 Definition of endpoint(s)

### 7.2.1.1 Number of confirmed UTIs

The number of confirmed UTIs for both the:

- Mean number of confirmed UTIs during the three months' intervention period, as compared to placebo.

and

- Mean number of confirmed UTIs during the three months' follow-up period, as compared to placebo.

will be analysed using the same methods as for the primary endpoint.

### 7.2.1.2 Time to first relapse of UTI

Time to first relapse of UTI will be defined as the time from delivery of intervention (i.e. start of intervention) to date of first confirmed UTI ((Confirm date – Intervention date) + 1).

Subjects with no UTI will be censored at last known date within the study period.

The time to first relapse will be analysed using Cox regression analysis and presented by Kaplan-Meier graphs.

### 7.2.1.3 Relapse rate

The relapse rate for both:

- Proportion of subjects (%) who experienced at least one confirmed UTI during three months from start of intervention, as compared to placebo.

and



CTC Project Code: 2017-149

- Proportion of subjects (%) who experienced at least one confirmed UTI during six months from start of intervention, as compared to placebo.

will be analysed using Chi-square test without continuity correction and presented using frequency tables.

### 7.2.2 Analysis safety endpoint(s)

### 7.2.2.1 Adverse events

Adverse events and SAEs will be recorded from start of IP intervention. Medical events occurring between screening and start of IP intervention will be reported separately.

### 7.2.3 Main analytical approach

The mean number of UTIs will be analysed using analysis of covariance with intervention, UTI history and age as independent variables. Sexual activity will only be used in the analysis if it is possible. No intervention by centre interaction will be possible to apply in this analysis. The estimated intervention difference will be presented by LSMeans and a 95% confidence interval. The time to first relapse of UTI will be analysed using Cox regression analysis and presented by Kaplan-Meier graphs.

### 7.2.4 Sensitivity analysis

No sensitivity analysis for secondary endpoint(s) will be performed.

### 7.2.5 Supplementary analyses

No supplementary analysis for secondary endpoint(s) will be performed.

### 7.2.6 Presentation

The p-values will be included in the summary tables.

### 7.3 Tertiary/Exploratory Endpoint(s) Analysis

No tertiary/exploratory analysis will be performed.

### 7.4 Discontinuation

Patients who discontinue from IMP treatment will be tabulated. The reason for discontinuation will be given. For discontinuation due to AE, the AEs will be given.

### 7.5 Other Analyses

No other analysis will be performed.

### 7.6 Interim Analysis

No interim analysis will be performed.



CTC Project Code: 2017-149

### **8 CHANGES FROM THE CSP**

The following have been adjusted regarding to the CSP:

- Sexual activity will only be used in the analysis if it is possible.
- The definition of confirmed and unique UTI's have been added.
- Specify the definition of compliance for PPS.
- Subjects who have been used prohibited medications, long term antibiotics or Hipex during the study will be excluded from PPS.
- Subjects not participated at visit 4 and 7 (3 month and 6 month) will not be included in the PPS population.



CTC Project Code: 2017-149

### 9 STATISTICAL DELIVERABLES

The following documents will be delivered:

- SAP
- Statistical analyses and summary tables



CTC Project Code: 2017-149

### 10 SOFTWARE

All statistical analyses will be performed using SAS Version 9.4 (SAS institute, Cary, NC).



CTC Project Code: 2017-149

### 11 APPROVAL

Issued by:

Fredrik Hansson, Director Biometrics

CTC Representative

03 SEP 2019
Date (dd-Mmm-yyyy)

Date (dd-Millin-yyyy)

Approved by:

Kerstin Nilsson, Clinical Research Manager BloGaia AB Representative

4 Sep 2019
Date (dd-Mmm-yyyy)



CTC Project Code: 2017-149

### 12 SUPPORTIVE DOCUMENTATION

### 12.1 Appendix 1. – List of Abbreviations

| AE ATC Anatomical-Therapeutic-Chemical BMI Body Mass Index CF Clean File Cfu Colony-forming units CRF Case Report Form CSP Clinical study protocol CTA Clinical Trial Agreement CV Curriculum Vitae DMP Data Management Plan DSM Deutsche Sammlung von Mikroorganismen DVP Data Validation Plan EERA European Economic Area FAS Full Analysis Set GI Gastro-intestinal ICF Informed Consent Form IEC Independent Ethics Committee IIP Investigational Product N N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis System SD Standard Deviation SDV Source Data Verification SDV Source Data Verification Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Enrolled subject Subject randomized Subject completed | Abbreviation of term | Explanation |
|---|---|---|
| BMI CF Clean File Cfu Colony-forming units CRF Case Report Form CSP Clinical study protocol CTA Clinical Trial Agreement CV Curriculum Vitae DMP Data Management Plan DSM Deutsche Sammlung von Mikroorganismen DVP Data Validation Plan eCRF Electronic Case Report Form EEA European Economic Area FAS Full Analysis Set GI Gastro-intestinal ICF Informed Consent Form IEC Independent Ethics Committee IIP Investigational Product N N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Event SAP Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Deprating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject Who has signed the Informed Consent Form (ICF) Screening failure Included subject Subject andomized but not completed Completed subject Subject completed both the intervention and the follow- | AE | Adverse Event |
| CF Cfu Cfu Colony-forming units CRF Case Report Form CSP Clinical study protocol CTA Clinical Trial Agreement CV Curriculum Vitae DMP Data Management Plan DSM Deutsche Sammlung von Mikroorganismen DVP Data Validation Plan ECRF Electronic Case Report Form EEA European Economic Area FAS Full Analysis Set GI Gastro-intestinal ICF Informed Consent Form IEC Independent Ethics Committee IIP Investigational Product N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Included subject Subject randomized Withdrawn subject Subject randomized Withdrawn subject Subject completed both the intervention and the follow- | ATC | Anatomical-Therapeutic-Chemical |
| cfu Colony-forming units CRF Case Report Form CSP Clinical study protocol CTA Clinical study protocol CTA Clinical Trial Agreement CV Curriculum Vitae DMP Data Management Plan DSM Deutsche Sammlung von Mikroorganismen DVP Data Validation Plan eCRF Electronic Case Report Form EEA European Economic Area FAS Full Analysis Set GI Gastro-intestinal ICF Informed Consent Form IEC Independent Ethics Committee IP Investigational Product N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAE Serious Adverse Reaction SAS Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary | вмі | Body Mass Index |
| CRF Case Report Form CSP Clinical study protocol CTA Clinical Trial Agreement CV Curriculum Vitae DMP Data Management Plan DSM Deutsche Sammlung von Mikroorganismen DVP Data Validation Plan EERA European Economic Area FAS Full Analysis Set GI Gastro-intestinal ICF Informed Consent Form IEC Independent Ethics Committee IP Investigational Product N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject on included Included subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | CF | Clean File |
| CSP Clinical study protocol CTA Clinical Trial Agreement CV Curriculum Vitae DMP Data Management Plan DSM Deutsche Sammlung von Mikroorganismen DVP Data Validation Plan ECRF Electronic Case Report Form EEA European Economic Area FAS Full Analysis Set GI Gastro-intestinal ICF Informed Consent Form IEC Independent Ethics Committee IP Investigational Product N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SDV Source Data Verification SDP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject on included Included subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | cfu | Colony-forming units |
| CTA Clinical Trial Agreement CV Curriculum Vitae DMP Data Management Plan DSM Deutsche Sammlung von Mikroorganismen DVP Data Validation Plan eCRF Electronic Case Report Form EEA European Economic Area FAS Full Analysis Set GI Gastro-intestinal ICF Informed Consent Form IEC Independent Ethics Committee IP Investigational Product N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SDV Source Data Verification SDP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject on included Withdrawn subject Subject randomized but not completed Completed subject | CRF | Case Report Form |
| CV Curriculum Vitae DMP Data Management Plan DSM Deutsche Sammlung von Mikroorganismen DVP Data Validation Plan ECRF Electronic Case Report Form EEA European Economic Area FAS Full Analysis Set GI Gastro-intestinal ICF Informed Consent Form IEC Independent Ethics Committee IP Investigational Product N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject to tincluded Included subject Subject randomized Withdrawn subject Subject randomized but not completed Completed subject | CSP | Clinical study protocol |
| DMP DSM Deutsche Sammlung von Mikroorganismen DVP Data Validation Plan ECRF Electronic Case Report Form EEA European Economic Area FAS Full Analysis Set Gl Gastro-intestinal ICF Informed Consent Form IEC Independent Ethics Committee IP Investigational Product N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SDV Source Data Verification SDP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject ont included Included subject Subject randomized Withdrawn subject Subject randomized but not completed Completed subject | СТА | Clinical Trial Agreement |
| DSM Deutsche Sammlung von Mikroorganismen DVP Data Validation Plan eCRF Electronic Case Report Form EEA European Economic Area FAS Full Analysis Set GI Gastro-intestinal ICF Informed Consent Form IEC Independent Ethics Committee IP Investigational Product N NMber MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject completed but not completed Completed subject | CV | Curriculum Vitae |
| DVP Data Validation Plan ECRF Electronic Case Report Form EEA European Economic Area FAS Full Analysis Set GI Gastro-intestinal ICF Informed Consent Form IEC Independent Ethics Committee IP Investigational Product N N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject completed both the intervention and the follow- | DMP | Data Management Plan |
| eCRF Electronic Case Report Form EEA European Economic Area FAS Full Analysis Set GI Gastro-intestinal ICF Informed Consent Form IEC Independent Ethics Committee IP Investigational Product N NUmber MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | DSM | Deutsche Sammlung von Mikroorganismen |
| EEA European Economic Area FAS Full Analysis Set GI Gastro-intestinal ICF Informed Consent Form IEC Independent Ethics Committee IIP Investigational Product N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Included subject Subject randomized Withdrawn subject Subject randomized Withdrawn subject Subject completed both the intervention and the follow- | | |
| FAS Full Analysis Set GI Gastro-intestinal ICF Informed Consent Form IEC Independent Ethics Committee IIP Investigational Product N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Uncluded subject Subject randomized Withdrawn subject Subject completed both the intervention and the follow- | | · |
| GI ICF Informed Consent Form IEC Independent Ethics Committee IP Investigational Product N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject rot included Included subject Subject randomized Withdrawn subject Subject completed both the intervention and the follow- | | |
| ICF Informed Consent Form IEC Independent Ethics Committee IP Investigational Product N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Withdrawn subject Subject randomized Withdrawn subject Subject completed both the intervention and the follow- | | • |
| IEC Independent Ethics Committee IP Investigational Product N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject completed both the intervention and the follow- | | |
| IP Investigational Product N Number MedDRA Medical Dictionary for Regulatory Affairs PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject completed both the intervention and the follow- | | |
| NNumberMedDRAMedical Dictionary for Regulatory AffairsPACProanthocyanidinPPSPer Protocol SetRCTRandomized Clinical TrialsSAESerious Adverse EventSAPStatistical Analysis PlanSARSerious Adverse ReactionSASStatistical Analysis SystemSDStandard DeviationSDVSource Data VerificationSOPStandard Operating ProceduresSUSARSuspected Unexpected Serious Adverse ReactionTMFTrial Master FileUTIUrinary Tract InfectionEnrolled subjectSubject who has signed the Informed Consent Form (ICF)Screening failureEnrolled subject not includedIncluded subjectSubject randomizedWithdrawn subjectSubject randomized but not completedCompleted subjectSubject completed both the intervention and the follow- | | |
| MedDRAMedical Dictionary for Regulatory AffairsPACProanthocyanidinPPSPer Protocol SetRCTRandomized Clinical TrialsSAESerious Adverse EventSAPStatistical Analysis PlanSARSerious Adverse ReactionSASStatistical Analysis SystemSDStandard DeviationSDVSource Data VerificationSOPStandard Operating ProceduresSUSARSuspected Unexpected Serious Adverse ReactionTMFTrial Master FileUTIUrinary Tract InfectionEnrolled subjectSubject who has signed the Informed Consent Form (ICF)Screening failureEnrolled subject not includedIncluded subjectSubject randomizedWithdrawn subjectSubject randomized but not completedCompleted subjectSubject completed both the intervention and the follow- | | _ |
| PAC Proanthocyanidin PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject completed both the intervention and the follow- | | |
| PPS Per Protocol Set RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | | |
| RCT Randomized Clinical Trials SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | | • |
| SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | | |
| SAP Statistical Analysis Plan SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject completed both the intervention and the follow- | | |
| SAR Serious Adverse Reaction SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | | |
| SAS Statistical Analysis System SD Standard Deviation SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | | |
| SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | | |
| SDV Source Data Verification SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | | |
| SOP Standard Operating Procedures SUSAR Suspected Unexpected Serious Adverse Reaction TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | | |
| SUSAR TMF Trial Master File UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Included subject Subject randomized Withdrawn subject Completed subject Subject completed both the intervention and the follow- | | |
| TMF UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Included subject Subject randomized Withdrawn subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | | |
| UTI Urinary Tract Infection Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | | · |
| Enrolled subject Subject who has signed the Informed Consent Form (ICF) Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Completed subject Subject completed both the intervention and the follow- | | |
| Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | 011 | Offinary fract infection |
| Screening failure Enrolled subject not included Included subject Subject randomized Withdrawn subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | Enrolled subject | Subject who has signed the Informed Consent Form (ICF) |
| Included subject Withdrawn subject Completed subject Subject randomized Subject randomized but not completed Subject completed both the intervention and the follow- | | |
| Withdrawn subject Subject randomized but not completed Completed subject Subject completed both the intervention and the follow- | _ | |
| Completed subject Subject completed both the intervention and the follow- | | • |
| | - | |
| | - | up periods |

### 12.2 Appendix 2. – Changes to Protocol-Planned Analyses

### 13 Demographic data

## 13.1 Demographic information

TABLE 14.1.1.1 SUMMARY OF DEMOGRAPHIC DATA AND OTHER BASELINE CHARACTERISTICS (FULL ANALYSIS SET)

| ABLE 14.1.1.1 SUMMARY OF L | I ABLE 14.1.1.1 SUMMAKY OF DEMOGRAPHIC DATA AND OTHER BASELINE CHARACTERISTICS (FULL ANALYSIS SET) | ERISTICS (FULL ) | ANALYSIS SET) | |
|---|---|---|---|---|
| | | Treatment A Treatment B (N=xx) | Treatment B (N=xx) | Total (N=xx) |
| Age (years) | n/nmiss | x/xx | x/xx | x/xx |
| | Mean (SD) | xx.x (x.x) | xx.x (x.x) | (x.x) x.xx |
| | Median (Min, Max) | xx.x (x, xx) | xx.x (x, xx) | xx.x (x, xx) |
| Weight (kg) | n/nmiss | x/xx | x/xx | x/xx |
| | Mean (SD) | xx.x (x.x) | xx.x (x.x) | xx.x (x.x) |
| | Median (Min, Max) | xx.x (x, xx) | xx.x (x, xx) | xx.x (x, xx) |
| Height (cm) | n/nmiss | x/xx | x/xx | x/xx |
| | Mean (SD) | xxx (x.x) | xx.x (x.x) | xx.x (x.x) |
| | Median (Min, Max) | xx.x (x, xx) | xx.x (x, xx) | xx.x (x, xx) |
| BM! (M2) | n/nmiss | x/xx | x/xx | x/xx |
| | Mean (SD) | xx.x (x.x) | xx.x (x.x) | xx.x (x.x) |
| | Median (Min, Max) | xx.x (x, xx) | xx.x (x, xx) | xx.x (x, xx) |

## 13.2 Medical/Surgical history

TABLE 14.1.4 MEDICAL HISTORY EVENTS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (FULL ANALYSIS SET)

| | Treatment A<br>N=xx | nt A | Treatment B<br>N=xx | nt B | Total<br>N=xx | |
|---|---|---|---|---|---|---|
| System organ class<br>Preferred term | (%)u | ٤ | u(%) | ٤ | u(%) | Ε |
| Total | (%xx)x | × | (%xx)x | × | (жж)х | × |
| Psychiatric disorders | (%xx)x | × | (%xx)x | × | (%xx)x | × |
| Anxiety | (%xx)x | × | (%xx)x | × | (%xx)x | × |
| Depression | (%xx)x | × | (%xx)x | × | (%xx)x | × |
| Insomnia | (%xx)x | × | (%xx)x | × | (%xx)x | × |
| Immune system disorders | (%xx)x | × | x(xx%) | × | (%xx)x | × |
| Hypersensitivity | (%xx)x | × | (%xx)x | × | (%xx)x | × |
| Seasonal allergy | (%xx)x | × | (%xx)x | × | (%xx)x | × |
| Metabolism and nutrition disorders | (%xx)x | × | x(xx)x | × | (%xx)x | × |
| Type 1 diabetes mellitus | (%xx)x | × | (%xx)x | × | (%xx)x | × |
| General disorders and administration site conditions | (%xx)x | × | x(xx)x | × | (%xx)x | × |
| Chronic fatigue syndrome | (%xx)x | × | (%xx)x | × | (%xx)x | × |
| Nervous system disorders | (%xx)x | × | (%xx)x | × | (%xx)x | × |
| Narcolepsy | (%xx)x | × | (%xx)x | × | (%xx)x | × |
| Reproductive system and breast disorders | (%xx)x | × | (%xx)x | × | (%xx)x | × |
| Premenstrual syndrome | (%xx)x | × | (%xx)x | × | (%xx)x | × |
| Respiratory, thoracic and mediastinal disorders | x(xx)x | × | (%xx)x | × | (%xx)x | × |
| Asthma | (%xx)x | × | (%xx)x | × | (%xx)x | × |
| Vascular disorders | (%xx)x | × | x(xx%) | × | x(xx%) | × |
| Hypertension | (%xx)x | × | (%xx)x | × | (%xx)x | × |

n, number of subjects; m, number of events. Percentages are based on the number of subjects in the full analysis set



## 13.3 Subject disposition and exposure

## TABLE 14.1.1.2 SUBJECT DISPOSITION

| | Treatment A | Treatment A Treatment B | Total |
|---|---|---|---|
| Screened subjects | X | XX | × |
| Subjects that entered the study | × | × | × |
| Withdrawn subjects | X | × | × |
| Completed subjects | X | X | × |
| Included in FAS | XX | × | × |
| Included in PPS* | X | × | × |
| Subjects at Screening | X | × | X |
| Subjects at Visit 2 | X | × | × |
| Subjects at Visit 3 | X | × | × |
| Subjects at Visit 4 | X | × | × |
| Subjects at Visit 5 | × | X | × |



## 13.4 CONCOMITANT MEDICATIONS

LISTING 16.2.5.2.1. CONCOMITANT MEDICATIONS, INDICATIONS (FULL ANALYSIS SET)

| Dosing<br>Frequency<br>per Interval | <u>^</u> | | As needed |
|---|---|---|---|
| Fr Fr | Daily | Daily | Asr |
| Route of<br>Administratio | Oral | Oral | Oral |
| Dose<br>Units A | mg Oral | mg | mg |
| Dose<br>Description | X | X | × |
| Dosing Medication Dose Dose Route of Frequency Class Code Category for Medication Description Units Administration per Interval | Medical/ surgical history | Medical/ surgical history | Medical/ surgical history |
| Medication<br>Class Code | XXX | XXX | XXX |
| Standardized Medication Name | 8 | × | 8 |
| | X | XX | XX |
| Reported Name of Drug,<br>Med, or Therapy | XK | XXK | XXK |
| Subject<br>dentifie<br>r for the Sequence<br>Study Number | X XXK | × | × |
| Subject<br>Identifie<br>r for the<br>Study | XX | XXX | XXX |
| Gender | Female | Female | Female |

### 13.5 Primary Endpoint: XXXX

TABLE 14.2xx XXXX (µg/l)

Variable

XXXX

| | | | Treatment A | Treatment B |
|---|---|---|---|---|
| Result Category | Visit Name | | | |
| Measured value | Visit 1 Baseline | z | × | X |
| | | Mean (SD) | (xxx) xx | (xxx) xx |
| | | Median (Min, Max) | xx (xx, xx) | xx (xx, xx) |
| | | 95% CI | xxtxx | xx;xx |
| | Visit 2 | z | × | × |
| | | Mean (SD) | (xxx) xx | (xxx) xx |
| | | Median (Min, Max) | xx (xx, xx) | xx (xx, xx) |
| | | 95% CI | xx;xx | xx;xx |
| Absolute change | Visit 2 | Z | × | × |
| trom baseline | | Mean (SD) | (xxx) xx | (xxx) xx |
| | | Median (Min, Max) | xx (xx, xx) | xx (xx, xx) |
| | | 95% CI | xx;xx | xx;xx |
| | | Between groups p-value (Wilcoxon) | 0.xxxx | 0.xxxx |
| | | Within group p-value (Wilcoxon) | 0.xxxx | 0.xxxx |
| Percent change from | Visit 2 | z | × | XX |
| baseline (%) | | Mean (SD) | xx (xxx) | xx (xxx) |
| | | Median (Min, Max) | xx (xx, xx) | xx (xx, xx) |
| | | 95% CI | xx;xx | xx;xx |
| | | Between groups p-value (Wilcoxon) | 0.xxxx | 0.xxxx |
| | | Within group p-value (Wilcoxon) | 0.xxxx | 0.xxxx |



# 13.6 Continuous variables measured over time

Variable

XXXXX

TABLE 14.2.xx Variables over time

| | | | Treatment A | Treatment B |
|---|---|---|---|---|
| Result Category | Visit Name | | | |
| Measured value | Visit 1 Baseline | Z | × | × |
| | | Mean (SD) | (xxx) xx | (xxx) xx |
| | | Median (Min, Max) | xx (xx, xx) | xx (xx, xx) |
| | | 95% CI | xx;xx | xx;xx |
| | XX | z | × | × |
| | | Mean (SD) | (xxx) xx | (xxx) xx |
| | | Median (Min, Max) | xx (xx, xx) | xx (xx, xx) |
| | | 95% CI | xx;xx | xx;xx |
| Absolute change | ×× | z | × | × |
| from baseline | | Mean (SD) | (xxx) xx | xx (xxx) |
| | | Median (Min, Max) | xx (xx, xx) | xx (xx, xx) |
| | | 95% CI | xx;xx | xx;xx |
| | | Between groups p-value (Wilcoxon) | 0.xxxx | 0.xxxx |
| | | Within group p-value (Wilcoxon) | 0.xxxx | 0.xxxx |
| Percent change from | XX | z | × | × |
| baseline (%) | | Mean (SD) | (xxx) xx | xx (xxx) |
| | | Median (Min, Max) | xx (xx, xx) | xx (xx, xx) |
| | | 95% CI | xxtxx | xx:xx |
| | | Between groups p-value (Wilcoxon) 0.xxxx | 0.xxxx | 0.xxxx |
| | | Within group p-value (Wilcoxon) | 0.xxxx | 0.xxxx |

# 13.7 Continuous variables measured at one occasion

TABLE 14.2.xx Variables at one occasion

| Treatment B | | × | (xxx) xx | xx (xx, xx) | xx:xx | 0.xxxx |
|---|---|---|---|---|---|---|
| Treatment A | | × | (xxx) xx | xx (xx, xx) | xx;xx | 0.xxxx |
| | | Z | Mean (SD) | Median (Min, Max) | 95% CI | Between groups p-value (Wilcoxon) 0.xxxx |
| | Visit Name | XXX | | | | |
| | Result Category Visit Name | Measured value | | | | |
| | Variable | XXXXX | | | | |



## 13.8 Categorical variables at different visits

TABLE 14.2.xx categorical variables over time

| | | Treatment A<br>(N=xx) | Treatment A Treatment B (N=xx) | Total (N=xx) |
|---|---|---|---|---|
| Prevalence of XXXXXXX visit x | No | (%xx) xx | (%xx) xx | (%xx) xx |
| | Yes | (%xx) xx | (%xx) xx | (%xx) xx |
| | Chi-Square p-value | | | 0.xxxx |

### 13.9 Adverse events

TABLE 14.3.1.1 OVERVIEW OF ADVERSE EVENTS, FAS

| | Treatment A<br>N=XX | Treatment B<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| | n(%) | u(%) | u(%) |
| Any AE | (%xx)x | x(xx%) | (%xx)x |
| Any SAE | (%xx)x | x(xx%) | (%xx)x |
| Any AE leading to<br>withdrawal | (%xx)x | ≭(xx%) | (%xx)x |
| Any AE leading to death | (%xx)x | x(xx%) | (%xx)x |
| Causality | | | |
| Not Related | (%xx)x | x(xx%) | (%xx)x |
| Possible | x(xx%) | x(xx%) | (%xx)x |
| Probable | (%xx)x | x(xx%) | (%xx)x |
| Severity | | | |
| PIIM | (%xx)x | ×(xx%) | (%xx)x |
| Moderate | (%xx)x | x(xx%) | (%xx)x |

n, number of subjects; m, number of subjects is number of events
Percentages are based on the number of subjects in the treatment period included in the full analysis set.
Adverse events that occurred during follow-up are omitted from summary.

TABLE 14.3.1.2 ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND PREFERRED TERM, FAS

Total N=XX

Treatment A Treatmen: B N=XX N=XX

| System organ class<br>Preferred term | n(%) | ٤ | n(%) | ٤ | m n(%) | Ε |
|--------------------------------------|--------|---|--------|---|--------|---|
| Gastrointestinal disorders | (%xx)x | > | x(xx%) | > | x(xx%) | > |
| Dry mouth | x(xx%) | > | (%xx)x | > | x(xx)x | > |
| Gingival blister | (%xx)x | > | x(xx%) | > | (%xx)x | > |
| Lip pain | (%xx)x | > | x(xx%) | > | x(xx)x | > |
| Nausea | (%xx)x | > | x(xx%) | > | x(xxx) | > |
| Infections and infestations | (%xx)x | > | x(xx%) | > | x(xx%) | > |
| Diarrhoea infectious | (%xx)x | > | x(xx%) | > | x(xx%) | > |
| Gastroenteritis viral | (%xx)x | > | x(xx%) | > | (%xx)x | > |
| Influenza | (%xx)x | > | x(xx%) | > | (%xx)x | > |
| Nasopharyngitis | (%xx)x | > | x(xx)x | > | x(xx)x | > |
| Nervous system disorders | (%xx)x | > | x(xx)x | > | (%xx)x | > |
| Dizziness | (%xx)x | > | (%xx)x | > | x(xx)x | > |

n, number of subjects; m, number of events
Percentages are based on the number of subjects in the treatment period included in the full analysis set.
Adverse events that occurred during follow-up are omitted from summary.

TABLE 14.3.1.3 ADVERSE EVENTS: SEVERITY AND RELATION, WITH PATIENT IDENTIFICATIONS, FAS

| | | | Mild | Mild<br>Related | Moderate<br><br>NR | Moderate<br>—-<br>Related | Total<br>II | Total<br>—<br>Related | Total<br>—<br>R+NR |
|---|---|---|---|---|---|---|---|---|---|
| Treatment A | Gastrointestinal disorders | Nausea | | (%xx) x | | | | (%xx) x | (%xx) x |
| (NXX) | | | | ** XXX | | | | | |
| | Infections and infestations Gastroenteritis viral | Gastroenteritis viral | | | (%xx) x | | (%x) x | | (%xx) x |
| | | | | | XXX | | | | |
| | | Nasopharyngitis | (%xx) x | | | | (%x) x | | (%xx) x |
| | | | XX | | | | | | |
| | Nervous system disorders | Dizziness | | (%xx) x | | | | (%xx) x | (%xx) x |
| | | | | XXX | | | | | |
| Treatment B | Gastrointestinal disorders Dry mouth | Dry mouth | | (%xx) x | | | | (%xx) x | (%xx) x |
| (var. | | | | XXX | | | | | |
| | | Gingival blister | | | | (%xx) x | | (%xx) x | (%xx) x |
| | | | | | | XXX | | | |
| | | Lip pain | (%xx) x | | | | × (%) | | (%xx) x |
| | | | XXX | | | | (%/YY) | | |
| | Infections and infestations Diarrhoea infectious | Diarrhoea infectious | | | (%)xx) x | | X (%) | | (%xx) x |
| | | | | | xxx | | (%//) | | |
| | | Influenza | (%xx) x | | | | × (%^^) | | (%xx) x |
| | | | XXX | | | | (0/00) | | |

\*\*: Subject randomisation number R: Related. NR: Not related. AEs judged as 'Possibly Related' or 'Problably Related' are grouped as 'Related'. Adverse events that occurred during follow-up are omitted from summary.

